CLINICAL TRIAL: NCT06967584
Title: Effects of Thoracic Kinesio Taping on Pulmonary Functions, Respiratory Muscle Strength and Functional Capacity in Patients With Hemiplegia
Brief Title: Kinesiotaping on HP Patients Pulmonary Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Çiçek Günday, Asst. Prof., Istinye University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1142025
Record Dates: First submitted 2025-04-19; First posted 2025-05-13 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Hemiplegic Patients; Hemiplegia
Keywords: Stroke; Kinesio taping; Chest Physiotherapy; Respiratory test
MeSH Terms: conditions — Hemiplegia; Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Taping group (Experimental)
  Interventions: Other: Kinesio Taping
- Sham Kinesio Taping group (Sham Comparator)
  Interventions: Other: Sham Kinesio Taping

INTERVENTIONS:
Other: Kinesio Taping — The Kinesio tape will be applied anteriorly and posteriorly along the subcostal region to facilitate the respiratory muscles. Anteriorly, an "I"-shaped Kinesio tape will be applied with the base anchored on the xiphoid process, stretched to 50-75% tension, applied only to the linea alba. The ends of the tape will be applied without tension toward the subcostal curvature. Posteriorly, a second "I"-shaped Kinesio tape will be applied. The base of the tape will be anchored on the spinous process of the 12th thoracic vertebra with 50-75% tension, and the tails will be applied without tension toward the ribs
  Arms: Kinesio Taping group
Other: Sham Kinesio Taping — The Kinesio tape will be applied anteriorly and posteriorly along the subcostal region but without tension
  Arms: Sham Kinesio Taping group

SUMMARY:
The aim of this study is to investigate whether thoracic kinesio taping contributes to the improvement of pulmonary function, the strengthening of respiratory muscles and the enhancement of overall physical ability in stroke patients with hemiplegia. To assess this, a randomized controlled trial will be conducted involving 30 patients aged between 45 and 80 years who have been diagnosed with hemiplegia resulting from a stroke. Participants will be randomly assigned to one of two groups: the Kinesio Taping Group (KTG) or the Sham Kinesio Taping Group (SKTG). The duration of the intervention will be four weeks. During this period, individuals in the KTG will receive thoracic kinesio taping in addition to standard rehabilitation care. In the SKTG, taping will be applied to the same thoracic area but without tension. Measurements will be obtained both before and after the intervention. These assessments will include pulmonary function tests (such as forced vital capacity and forced expiratory volume), evaluations of respiratory muscle strength (specifically maximum inspiratory pressure), and assessments of functional capacity.

DETAILED DESCRIPTION:
Hemiplegia, a condition commonly occurring after a stroke, results in paralysis or significant weakness on one side of the body. Although it is primarily recognized for limiting movement in the limbs, hemiplegia can also profoundly affect respiratory function. Many individuals with hemiplegia experience compromised respiratory performance, which can negatively impact overall health, delay recovery, and reduce quality of life. When a stroke affects brain regions responsible for motor control, it may also impair the muscles involved in breathing. Consequently, individuals with hemiplegia often present with weakened respiratory muscles, restricted thoracic mobility, and diminished lung function. These impairments can lead to insufficient oxygen intake, increased susceptibility to respiratory infections such as pneumonia, and prolonged hospitalization. In addition to muscle weakness, patients may develop stiffness in the chest wall and diaphragm, which limits thoracic expansion during inhalation. This restriction can reduce lung capacity and increase the effort required for breathing. Over time, decreased movement in the thoracic region may result in muscle fibrosis and further loss of flexibility. These changes contribute to symptoms such as dyspnea, fatigue, and reduced functional capacity in daily activities. Furthermore, malnutrition-commonly observed in individuals with neurological conditions like stroke-can exacerbate respiratory muscle weakness and increase the risk of respiratory failure. The interplay between poor nutritional status, weakened respiratory muscles, and compromised lung function may create a detrimental cycle that hinders recovery. To improve pulmonary function in patients with hemiplegia, thoracic kinesio taping may be a promising method. This technique involves applying elastic therapeutic tape to the thoracic region to support muscular function, improve posture, enhance breathing mechanics, and increase proprioceptive awareness.

The present study aims to determine whether thoracic kinesio taping can enhance pulmonary function (i.e., lung performance), strengthen respiratory muscles (particularly those involved in inspiration), and improve overall physical capacity in stroke patients with hemiplegia. To evaluate this, a randomized controlled trial will be conducted involving 30 patients between the ages of 45 and 80 who have been diagnosed with hemiplegia resulting from a stroke. All participants will be medically stable and will have experienced a stroke within the previous six months. Patients with significant cardiac or neurological comorbidities, psychiatric conditions impairing communication, or dermatological sensitivities will be excluded to ensure safety and data integrity.

The intervention will span four weeks. During this period, participants will receive thoracic kinesio taping in addition to standard rehabilitation care. In the control group, sham taping will be applied to the same thoracic region without tension. Assessments will be performed before and after the intervention. These will include pulmonary function tests (e.g., forced vital capacity and forced expiratory volume), measurements of respiratory muscle strength (specifically maximum inspiratory pressure, or MIP), and evaluations of functional capacity. It is anticipated that an improvement in MIP may be observed, suggesting a strengthening of inspiratory muscles due to the intervention. No significant changes are expected in maximum expiratory pressure (MEP), which assesses expiratory muscle strength. Any observed improvements in respiratory parameters and daily functional abilities would support the efficacy of thoracic kinesio taping as a supplementary tool in stroke rehabilitation.

This study holds significance by addressing a frequently overlooked component of stroke recovery: respiratory health. Identifying effective strategies to support pulmonary function may enhance recovery outcomes, reduce complications, and promote greater independence in daily life. The results of this study may also inform the development of more comprehensive rehabilitation protocols for individuals with hemiplegia.

ELIGIBILITY:
Inclusion Criteria:

* The patients with stroke diagnosis by a neurologist
* 45-80 years old
* Participating to the study in a voluntary basis.
* Patients with clinical setting
* Patient diagnosed at lest stroke attack within 6 months
* They are Medically stable situation

Exclusion Criteria:

* Any Other neurological or orthopedic problems that will affect function other than Stroke
* Patients having unstable
* Severe heart diseases like heart failure, unstable hypertension, previous angina pectoris or myocardial infarction
* Skin sensitivity against kinesio tape
* Lesion or incision in the area of kinesio tape application
* Use of analgesics during study period .
* Mental and cognitive disorders that would affect cooperation.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | Through study completion, an average of 1 month
  Pulmonary function testing will be performed in a sitting position using a portable spirometer according to American Thoracic Society guidelines. Spirometry is a standard pulmonary function test used to assess how effectively the lungs are operating. The test will calculate FVC (The volume delivered during an expiration made as forcefully and completely as possible starting from full inspiration)
Forced Expiratory Volume in the first second (FEV1) | Through study completion, an average of 1 month
  Pulmonary function testing will be performed in a sitting position using a portable spirometer according to American Thoracic Society guidelines. Spirometry is a standard pulmonary function test used to assess how effectively the lungs are operating. The test will calculate FEV1 (The volume delivered in the first second of a FVC maneuver.)
Peak Expiratory Flow (PEF) | Through study completion, an average of 1 month
  Pulmonary function testing will be performed in a sitting position using a portable spirometer according to American Thoracic Society guidelines. Spirometry is a standard pulmonary function test used to assess how effectively the lungs are operating. The test will calculate PEF (The highest forced expiratory flow measured with a peak flow meter. In other word, this measures the maximum speed at which the patient can exhale air.)
Respiratory Muscle Strength | Through study completion, an average of 1 month
  Respiratory muscle strength, including maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP), will be evaluated using an electronic pressure transducer (MicroRPM; Micro Medical Ltd., Kent, United Kingdom). For the MIP measurement, the patient will be seated comfortably. Following a maximal exhalation, the nose will be occluded using a nasal clip, and a maximal inhalation will be performed through a mouthpiece. For the MEP measurement, after a maximal inhalation in the same seated position, the nose will again be closed with a clip, and a maximal exhalation will be carried out through the mouthpiece. Each measurement will be repeated three times, and the highest value will be recorded. Assessments will be performed twice: once at baseline and once at the end of the approximately one-month intervention period.
Functional Capacity | Through study completion, an average of 1 month
  Functional capacity will be assessed using the Functional Bridge Test (FBT). In this test, the patient lies in a supine position on a bed and performs a bridge movement, which involves lifting the hips and extending the trunk against gravity, thereby engaging the hip and trunk extensor muscles. This maneuver is intended to evaluate the postural control function of the proximal lower-extremity and trunk muscles, which are essential for bed mobility. The test is graded on a four-point scale to assess functional capacity:
  Grade 1: Difficulty initiating lift-off Grade 2: Insufficient hip elevation Grade 3: Slightly insufficient hip elevation Grade 4: Sufficient hip elevation Assessments will be conducted twice: once at baseline and once at the end of the one-month intervention period.

SECONDARY OUTCOMES:
Symptoms- Dyspnea, Fatigue, pain, cough and sputum | Through study completion, an average of 1 month
  The patient's pain intensity, severity of dyspnea, and cough severity will be evaluated using the Visual Analog Scale (VAS), a tool that helps assess the intensity of sensations such as pain. The VAS consists of a straight line, with one end indicating no pain "0" and the other end representing the worst pain imaginable "10", allowing patients to mark a point that corresponds to their experience. Additionally, the presence of sputum will be evaluated through patient questioning to further assess respiratory symptoms.
Functional Independence Measure | Through study completion, an average of 1 month
  The Functional Independence Measure (FIM) is one of the most highly recommended tools for assessing functional recovery in stroke patients. This tool is considered reliable and has been proven to possess high validity for measuring the functional outcomes of stroke patients. FIM consists of 18 items related to daily activities, with a total score ranging from 18 to 126. Each item is rated on a 7-point scale, ranging from 1 (completely dependent) to 7 (independent), based on the level of independence. A total score of ≤108 indicates the need for assistance or limitations in activities.
Muscle Strength | Through study completion, an average of 1 month
  The muscle strength will assess by using the hand held dynamometer. Muscle strength of shoulder flexors, abductors, elbow flexors, hip flexors, hip extensors and knee extensors will be evaluated.
Grip Strength | Through study completion, an average of 1 month
  JAMAR hand dynamometer will be used to evaluate grip strength. During the grip strength assessment, subjects will instruct to position their hand on their thigh with adduct and neutrally rotated shoulders. The arm being test had the elbow flexed to 90 degrees, while the forearm, wrist, and fingers maintained neutral positions
Muscle Tone | Through study completion, an average of 1 month
  The Muscle Tone will be measured by using Modified Ashworth Scale. Modified Ashworth Scale tool used to measure the increase of muscle tone in stroke patients. Ashworth Scale as a method of grading spasticity while working with stroke. The original Ashworth scale was a 5 point numerical scale that graded spasticity from 0 to 4, with 0 being no resistance and 4 being a limb rigid in flexion or extension.

CONTACTS AND LOCATIONS:
Overall Officials: Roya Soltanalizadeh, Specialist, Study Chair — Istinye University; Yunus Emre Tütüneken, Pt.MSc.PhD, Study Chair — Istinye University
Locations (1):
- İstinye University Bahçeşehir Liv Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No